CLINICAL TRIAL: NCT04619459
Title: The Effect of Kangaroo Mother Care Applied to the Healthy Newborns in the Early Postpartum Period on Breastfeeding: Randomized Controlled Study
Brief Title: The Effect of Kangaroo Mother Care Applied to the Healthy Newborns on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sevda KORKUT ÖKSÜZ, Research Assistant, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AhiEvranEDU
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Breastfeeding; Kangaroo Mother Care; Breastfeeding, Exclusive
Keywords: Kangaroo Mother Care; Breastfeeding; Postpartum Period; Term Newborn; Midwifery
MeSH Terms: conditions — Breast Feeding | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborns receiving Kangaroo Mother Care (KMC) (Experimental): The newborns' diapers were tied, their caps put on and then they were positioned on their mother's naked chest for KMC. At Minute 5, the newborns' Apgar scores were assessed and recorded during KMC. The newborn's examination and injections (Hepatitis-B and K vit) were postponed until the first breastfeeding took place. A pediatrician performed a detailed examination of the newborns under the radiant infant warmer after the first breastfeeding. Following the examination, the newborn was positioned on the mother's breast for KMC. During this KMC, the newborn was administered 1 mg K vitamin in the right leg and 0.5 ml Hepatitis-B vaccine in the left leg via intramuscular injections. The KMC session was continued for 3 hours. Care attempt of mothers such as episiotomy repair was taken that the position of KMC.
  Interventions: Other: Kangaroo Mother Care (KMC)
- Newborns receiving standard postpartum care (SPC): (No Intervention): He received the standard care of the hospital. KMC not applied.

INTERVENTIONS:
Other: Kangaroo Mother Care (KMC) — Kangaroo mother care is a method of care of infants. The method involves infants being carried, usually by the mother, with skin-to-skin contact. Kangaroo mother care (KMC). early after delivery have better success at breastfeeding and achieve this success sooner. In this method The newborns' diapers were tied, their caps put on and then they were positioned on their mother's naked chest for KMC. The KMC session was continued for 3 hours.
  Arms: Newborns receiving Kangaroo Mother Care (KMC)

SUMMARY:
This study aims to determine the effect of kangaroo mother care (KMC) applied to the healthy newborns in the early postpartum period on breastfeeding.

The results of the study are expected to contribute to promoting the practice of KMC in an effort to encourage breastfeeding not only in Turkey's hospitals but also in other developing countries where practices that negatively affect breastfeeding are prevalent.

The hypotheses of the study were determined as: Infants administered KMC start to breastfeed sooner (H1), breastfeed more frequently (H2), breastfeed for longer periods (H3), are more successful at breastfeeding (H4) than infants receiving standard postpartum care (SPC).

DETAILED DESCRIPTION:
Setting: The study was conducted over the period June 1 - August 25, 2016 as randomized controlled experimental research at a Training and Research Hospital in Istanbul, Turkey.

Participants: The participants were 112 healthy mothers and their babies; the women were between the ages 18-42, had delivered normal vaginal birth between gestational weeks 38-40, met the sample inclusion criteria and consented to be a part of the study. Instrumental vaginal deliveries were excluded from this study.

The sample selection criteria were determined as: normal delivery, healthy mother and child, newborn being at term (in the 38th-42nd week), with a birthweight of 2500-4000 gr. The inclusion criteria were determined as: no serious case of asphyxiation in the newborn, an APGAR score of at least 7 at Minute 1 and Minute 5, no health problem in the newborn to prevent it from breastfeeding (e.g., cleft palate, harelip, esophageal atresia).

Sample and randomization: The researcher met with the mothers who fulfilled the selection criteria prior to the birth and briefly informed them of the scope and content of the study, asking them if they wished to participate. At this stage, participation was proposed to 119 mothers. Of these, 112 mothers and their babies were randomized into two groups with 56 in the study group (KMC) and 56 in the control group (SPC). A computerized randomization method was used for implementing the random selection. The newborns that exhibited a health issue following the birth were excluded from the study. In their place, the same randomization method was used until 56 cases were defined. The number of newborns held outside the scope of the study after birth was 5 in the study group and 2 in the control group.

Power analysis was performed using the G*Power (v3.1.9) program in order to determine the number in the sample. Sample size was determined on the basis of the infants' breastfeeding scores obtained on LATCH. It was foreseen that a unit of difference in LATCH scores between groups would be clinically significant. In a study by Yenal et al., when the LATCH mean score and standard deviation were accepted as a reference for control group data, effect size was calculated as d=0.566. It was calculated that at least 51 individuals would have to be included in the groups, a total of 102, to realize the effect level of α=0.05 at a power of 80%. Taking into consideration possible losses, it was decided that the groups would each comprise at least 56, meaning a total of 112 individuals.

Data collection: The study data were collected in line with the literature using the Data Collection Form developed by researchers. The infants' suckling skills were assessed with the "LATCH Breastfeeding Assessment Tool" developed in 1994 by Jensen et al.

Consent: Permission for conduct of the study was obtained from the hospital and the ethics committee (10840098-604.01.01-E.1108). At the same time, prior to the start of the study, the mothers were informed about the purpose and methodology of the research and the mothers agreeing to participate were asked to sign a written Subject Informed Consent Form.

Data analysis: The NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah, USA) program was used in the statistical analysis. In the evaluation of the study data, besides descriptive statistical methods (means, standard deviation, median, frequency and percentages), the Shapiro-Wilk test and box plot graphs were employed in testing normality. The Independent Samples T Test was used to analyze two groups of quantitative data displaying normal distribution such as the newborns' weight, height, head circumference, number of breastfeedings received, mother's age. The Mann-Whitney U test was used in the case of variables not showing normal distribution, such as the newborns' APGAR scores at Minutes 1 and 5, the first interaction of the mother with her infant, the first time of breastfeeding, the number of breastfeedings in the first 3 hours and their duration. The comparison of qualitative data such as the infants' gender, the mother's educational status, the status of being breastfed in the first half-hour and hour was undertaken with Pearson's Chi Square while the Fisher-Freeman-Halton test was used to compare the mothers' eagerness to breastfeed. The results were analyzed at a confidence interval of 95% with significance expressed at a level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers
* The women were between the ages 18-42,
* Had delivered normal vaginal birth
* Between gestational weeks 38-40
* Consented to be a part of the study
* Newborn being at term (in the 38th-42nd week), with a birthweight of 2500-4000 gr.
* No serious case of asphyxiation in the newborn,
* APGAR score of at least 7 at Minute 1 and Minute 5,
* No health problem in the newborn to prevent it from breastfeeding

Exclusion Criteria:

* Instrumental vaginal deliveries
* Cesarean deliveries

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the women were between the ages 18-42, had delivered normal vaginal birth
Enrollment: 112 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding Assessment Tool | It was used in both groups before the first breastfeeding.
  The infants' suckling skills were assessed with this scale. The infants' suckling skills were assessed with the "LATCH Breastfeeding Assessment Tool" developed in 1994 by Jensen et al. and for which the validity and reliability testing of the Turkish version had been conducted by Yenal and Okumuş in 2003. The LATCH instrument comprises five parameters (Latch on breast, Audible swallowing, Type of nipple, Comfort breast/nipple, Hold/help) on which each item is assessed on the basis of 0-2. The highest possible score on the scale is 10; the lowest is 0.
LATCH Breastfeeding Assessment Tool | After 24 hours the sucking ability of both groups was evaluated.
  The infants' suckling skills were assessed with this scale. The infants' suckling skills were assessed with the "LATCH Breastfeeding Assessment Tool" developed in 1994 by Jensen et al. and for which the validity and reliability testing of the Turkish version had been conducted by Yenal and Okumuş in 2003. The LATCH instrument comprises five parameters (Latch on breast, Audible swallowing, Type of nipple, Comfort breast/nipple, Hold/help) on which each item is assessed on the basis of 0-2. The highest possible score on the scale is 10; the lowest is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda K Öksüz, R.A, Principal Investigator — Ahi Evran University Faculty of Health Sciences
Locations (1):
- Sevda Korkut Öksüz, Kırşehir, Bagbası, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I did not find it appropriate to share it.

REFERENCES:
- [Background] Inal S, Aydin Y, Canbulat N. Factors associated with breastfeeding initiation time in a baby-friendly hospital in Istanbul. Appl Nurs Res. 2016 Nov;32:26-29. doi: 10.1016/j.apnr.2016.03.008. Epub 2016 Apr 1. PMID 27969039
- [Background] Thukral A, Sankar MJ, Agarwal R, Gupta N, Deorari AK, Paul VK. Early skin-to-skin contact and breast-feeding behavior in term neonates: a randomized controlled trial. Neonatology. 2012;102(2):114-9. doi: 10.1159/000337839. Epub 2012 Jun 14. PMID 22699241
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Schiff DM, Wachman EM, Philipp B, Joseph K, Shrestha H, Taveras EM, Parker MGK. Examination of Hospital, Maternal, and Infant Characteristics Associated with Breastfeeding Initiation and Continuation Among Opioid-Exposed Mother-Infant Dyads. Breastfeed Med. 2018 May;13(4):266-274. doi: 10.1089/bfm.2017.0172. Epub 2018 Apr 9. PMID 29630387
- [Background] Aghdas K, Talat K, Sepideh B. Effect of immediate and continuous mother-infant skin-to-skin contact on breastfeeding self-efficacy of primiparous women: a randomised control trial. Women Birth. 2014 Mar;27(1):37-40. doi: 10.1016/j.wombi.2013.09.004. Epub 2013 Nov 9. PMID 24216342
- [Background] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Derived] Oksuz SK, Inal S. The effect of kangaroo mother care applied to the healthy newborns in the early postpartum period on breastfeeding: A randomized controlled trial. J Pak Med Assoc. 2021 Sep;71(9):2124-2129. doi: 10.47391/JPMA.376. PMID 34580499